CLINICAL TRIAL: NCT05279716
Title: Safety and Efficacy Study in NTG, POAG, Glaucoma Suspect, Ocular Hypertension Patients With Diagnosed Prostaglandin Associated Peri-orbitopathy Switching From Preserved Prostaglandin Analogues Monotherapy to Omidenepag Isopropyl
Brief Title: Study in Prostaglandin Associated Peri-orbitopathy Switching From Prostaglandin Monotherapy to Omidenepag Isopropyl
Acronym: NOPAPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Santen Pharmaceutical Asia Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO-PAPS-Study
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Normal Tension Glaucoma; Primary Open-angle Glaucoma; Glaucoma, Suspect; Ocular Hypertension
Keywords: prostaglandin associated peri-orbitopathy(PAPS)
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- omidenepag isopropyl 0.02mg (Experimental): Instill 1 drop of Eybelis ophthalmic solution 0.002% once a day into the affected eye.
  Interventions: Drug: Eybelis ophthalmic solution 0.002%

INTERVENTIONS:
Drug: Eybelis ophthalmic solution 0.002% — Ophthalmic eye drop
  Other Names: Omidenepag isopropyl ophthalmic solution

SUMMARY:
This study is for patients have been using prostaglandin analogue eye drops with a preservative for 3 months or more and have been diagnosed with prostaglandin-associated peri-orbital disease.

the investigators would like to confirm the real world evidence(RWE) of safety and efficacy after changing to Eybelis ophthalmic solution 0.002%.

DETAILED DESCRIPTION:
This clinical trial is a single-arm, multicenter, prospective clinical trial, in which participants have consented to participate in the clinical trial are sequentially registered and proceeded.

The participant's participation period is a total of 24 weeks after the 4-week wash-out period, and according to the visit schedule, tests according to medical procedures are conducted at Screening, Baseline, 6, 12, 18, and 24 weeks to collect data on safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 19 and 79 years of age.
2. Normal Tension Glaucoma, Primary open-angle glaucoma, Glaucoma suspect and Ocular hypertension patients.
3. Patients who have received prostaglandin analogue (PGA) eye drops with preservatives for at least 3 months from the date of consent.
4. Patients diagnosed with prostaglandin associated peri-orbitopathy due to the use of Prostaglandin analogue (PGA) eye drops with preservatives.

   * DUES (Deepening of Upper Eyelid Sulcus)
   * FLEB (Flattening of Lower Eyelid Bag)
   * Upper eyelid ptosis
   * Periorbital hyperpigmentation
   * Ciliary hypertrichosis
5. Those who have agreed in writing to participate in this clinical trial.

Exclusion Criteria:

1. Patients with glaucoma caused by secondary causes such as pseudo-exfoliative glaucoma and pigment dispersion syndrome
2. Patients with intraocular pressure greater than 34 mmHg
3. Patients with severe visual impairment (Mean deviation -20dB or more)
4. History of eye surgery within 6 months from the date of consent (Corneal refractive surgery or intraocular surgery including LASIK and LASEK that affect the condition of the ocular surface)
5. Patients with severe dry eyes (those receiving or in need of drug treatment), those with eye allergies, infections, or inflammatory diseases
6. Those who are using systemic or eye steroids (except for topical skin)
7. Those who are using eye drops for the treatment of glaucoma other than Prostaglandin analogues eye drops with preservatives
8. Pregnant or lactating women
9. Those with hypersensitivity to anesthetic eye drops, fluorescein, or research drugs
10. Those who need to wear contact lenses during the clinical trial period
11. Artificial lens eye (pseudophakia) or aphakic eye (aphakia)
12. Periocular trauma, surgical history, or thyroid orbitopathy affecting the evaluation of prostaglandin associated peri-orbitopathy
13. Other clinical investigators judged to be inappropriate to participate in clinical trials

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-08 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of DUES(Deepening of Upper Eyelid Sulcus) | 24 weeks
  Primary efficacy parameter in prostaglandin associated peri-orbitopathy diseases at 24 weeks compared to baseline.
  -DUES (Deepening of Upper Eyelid Sulcus) Evaluate based on the following criteria.
  Grading is evaluated from 0 to 4 points. grade 0 = none; grade 1 = trace, barely visible; grade 2 = mild; grade 3 = moderate, easily detected; grade 4 = severe;

SECONDARY OUTCOMES:
Improvement rate of FLEB (Flattening of Lower Eyelid Bag) | 24 weeks
  second efficacy parameter in prostaglandin associated peri-orbitopathy diseases at 24 weeks compared to baseline.
  Facial photos, including eyebrows and lower eyelids, are taken by the investigator with the same digital camera and without flash in the same room conditions.
  When registering participants, the principal investigator of the conducting institution evaluates and registers participants, and the final evaluation is evaluated by three independent evaluators by randomly arranging the pictures taken during the visit so that the order of the visit is unknown.
Improvement rate of Upper eyelid ptosis in prostaglandin-associated peri-orbitopathy | 24 weeks
  second efficacy parameter in prostaglandin associated peri-orbitopathy diseases at 24 weeks compared to baseline.
  -Upper eyelid ptosis Margin reflex distance (MRD) is measured, and MRD 1 and MRD 2 are measured, respectively.
  This is measured to evaluate the palpebral fissure height.
  Grading is evaluated by the difference between the values of MRD 1 and MRD 2. mild = less than 2 mm; moderate = more than 2 mm and less than 4 mm; severe = more than 4 mm;
Improvement rate of Periorbital hyperpigmentation in prostaglandin-associated peri-orbitopathy | 24 weeks
  second efficacy parameter in prostaglandin associated peri-orbitopathy diseases at 24 weeks compared to baseline.
  -Periorbital hyperpigmentation Periorbital hyperpigmentation around the eyes is evaluated compared to the surrounding skin.
  Grading is evaluated from 0 to 4 points. grade 0 = skin color comparable to other facial skin areas; grade 1 = faint pigmentation of infraorbital fold; grade 2 = pigmentation more pronounced; grade 3 = deep dark color, all four lids involved; grade 4 = grade 3+ pigmentation spreading beyond infraorbital fold;
Improvement rate of Ciliary hypertrichosis in prostaglandin-associated peri-orbitopathy | 24 weeks
  second efficacy parameter in prostaglandin associated peri-orbitopathy diseases at 24 weeks compared to baseline.
  Facial photos, including eyebrows and lower eyelids, are taken by the investigator with the same digital camera and without flash in the same room conditions.
  When registering participants, the principal investigator of the conducting institution evaluates and registers participants, and the final evaluation is evaluated by three independent evaluators by randomly arranging the pictures taken during the visit so that the order of the visit is unknown.
Changes in intraocular pressure (IOP) | 24 weeks
  second efficacy parameter in intraocular pressure at 24 weeks compared to baseline.
Response rate of changes in intraocular pressure (IOP) | 24 weeks
  second efficacy parameter in Response rate of changes in intraocular pressure at 24 weeks compared to baseline.
Expression rate, number and change of Conjunctival Hyperemia | 24 weeks
  - Conjunctival Hyperemia Conjunctival Hyperemia is performed according to the evaluation criteria of the Japanese Ocular Allergy Society (JOAS).
  Grading is evaluated from 0 to 3 points. Grade 0 = No vasodilation; Grade 1= Some vessel vasodilation; Grade 2 = Excessive vessel vasodilation; Grade 3 = Overall vasodilation;
Expression rate, number and change of Macular Edema | 24 weeks
  -Macular Edema
  Inspect with Optical Coherence Tomography.
  Clinically significant macular edema in the following cases evaluate.
  * Thickening of the retina at or within 500 μm of the center of the macula.
  * Hard exudates at or within 500 μm of the center of the macula that associated with thickening of adjacent retina (which may lie more than 500 μm from the center of the macula).
  * A zone or zones of retinal thickening 1 disc area or larger, any part of which is within 1 disc diameter of the center of the macula
Expression rate, number and change of Cystoid Macular Edema | 24 weeks
  -Cystoid Macular Edema
  Inspect with Optical Coherence Tomography. CME I = cysts less than 30% macular thickness; CME II = cysts between 30% and 60% of macular thickness; CME III = cysts between 60% and 90% of macular thickness; CME IV = cysts became more than 90% of the macular thickness;
Expression rate, number and change of Endothelial Cell Count | 24 weeks
  -Endothelial Cell Count
  Measure with a specular microscope and check CD (Cell Density, cells/mm^2), CV (Coefficient of Variation), HEX (Hexagonality, %), NUM (number excluding incorrect count cells when counting cells) do.
Expression rate, number and change of Central Corneal Thickness | 24 weeks
  -Central Cornea Thickness
  After eye drop anesthesia, it is measured with an Ultrasonic Pachymeter(μm).

CONTACTS AND LOCATIONS:
Overall Officials: Munseok Kook, Principal Investigator — Asan Medical Center
Locations (8):
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Kim's Eye Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul ST. Mary's Hospital, Seoul
  - Severance Hospital, Seoul